CLINICAL TRIAL: NCT03133910
Title: Pharmacokinetics and Pharmacodynamics of Ceftazidime in Pediatric ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-679
Record Dates: First submitted 2017-03-09; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Sepsis
Keywords: Pharmacokinetics; Ceftazidime
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mortality benefit has been proven with early antibiotic administration in sepsis. Antimicrobial therapy should be based on early achievement of effective drug concentrations by optimizing the pharmacokinetic/pharmacodynamics of individual drugs. Optimal dosing in the critically ill patient can be challenging with the rapidly changing physiology of sepsis during the first days of hospitalization with capillary leak, fluid overload, changes in cardiac output, and alterations renal clearance. Ceftazidime is the preferred beta-lactam for empiric treatment of sepsis at Lurie Children's Hospital because of its anti-pseudomonal and anti-enteric bacilli coverage, however, the majority of pharmacokinetic data currently published in pediatrics does not include Intensive Care Unit (ICU) patients. Adult pharmacokinetic/pharmacodynamics data suggest that critically ill adults with high level of illness severity may benefit from continuous or extended infusion beta lactam therapy to optimize the therapeutic concentration particularly for pathogens that are relatively resistant to beta-lactams. Understanding the changing pharmacokinetic/pharmacodynamics of ceftazidime with the progression of illness in the ICU may help determine if current dosing regimens are adequate to maintain appropriate drug concentrations to optimize antimicrobial treatment.

DETAILED DESCRIPTION:
Severe sepsis continues to be a leading cause of admission and death in the pediatric critical care population. Mortality benefit has been proven with early antibiotic administration. Optimal antimicrobial therapy should be based on early achievement of effective drug concentrations by optimizing the pharmacokinetic/pharmacodynamics of individual drugs. Ceftazidime is the preferred beta-lactam for empiric treatment of sepsis at Lurie Children's Hospital because of its anti-pseudomonal and anti-enteric bacilli coverage, however, the majority of pharmacokinetic data currently published in pediatrics does not include ICU patients. For beta-lactams like ceftazidime, the time that free (nonprotein bound) drug concentration remains above the minimum inhibitory concentration (MIC) of the bacteria (t>MIC) best defines the bacteriostatic and bactericidal activity. Based on previous animal studies and subsequent clinical studies, beta-lactams require about 50% t>MIC. Adult pharmacokinetic/pharmacodynamics data suggest that critically ill adults with high level of illness severity may benefit from continuous or extended infusion beta lactam therapy to optimize time above MIC particularly for pathogens that are relatively resistant to beta-lactams. Positive outcome results using extended infusion have been found with respect to mortality benefit, clinical cure, reduced length of stay, and increased ventilator free days. It is likely that because children experience changes in physiology with critical illness likely leading to alteration in antibiotic clearance, additional data are needed to determine if our current dosing strategies are achieving optimal antimicrobial exposure. Understanding the changing pharmacokinetic/pharmacodynamics of ceftazidime with the progression of illness in the ICU may help determine if current dosing regimens are adequate to maintain appropriate t>MIC. In this study all patients between the ages of 2 months and 18 years admitted to the Pediatric Intensive Care Unit/ Cardiac Intensive Care Unit (PICU/CICU) who will receive ceftazidime for empiric or definitive antimicrobial therapy with an expected duration of greater than or equal to 48 hours who meet inclusion criteria will be enrolled in this prospective, non-interventional, pharmacokinetic study. Sampling of serum to determine concentrations will occur around ceftazidime doses during the first 48 hours after admission or onset of hospital associated illness, with additional sampling up to 7 days if antibiotic use continues. Using a traditional FDA-approved dosing regimen (50 mg q 8hr with maximum dosing of 6g/d), samples will be drawn following the 2nd or 3rd dose of Ceftazidime received by the patient at times: 0 min (predose), 30 min, 1 hour, and 4 hours following dose. During the second 24 hours of therapy, one sample will be drawn between hours 2 and 4 post dose and if therapy continues additional samples will be drawn daily between hours 2 and 4 post dose up to 7 days. Additional information will be collected to better assess volumes of distribution, drug clearance, kidney function, and cardiac output to determine patient covariates that may help delineate which patient populations associated with altered ceftazidime exposure. Population pharmacokinetic modeling will be performed and various regimens will be simulated to identify optimal dosing.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to pediatric or cardiac intensive care unit
* Between the ages of 2 month to 18 years
* Receiving ceftazidime for an anticipated course of greater than or equal to 48 hours
* Central venous or arterial access for blood sampling

Exclusion Criteria:

* Less than 2 months or greater than 18 years
* Anticipated need for renal replacement therapy or ECMO
* History of chronic kidney disease greater than stage 1
* Inadequate access for blood draws

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the ages of 2 months and 18 years admitted to the PICU/CICU who will receive ceftazidime for empiric or definitive antimicrobial therapy with an expected duration of greater than or equal to 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Duration of time that antibiotic concentration is above the minimum inhibitory concentration (T>MIC) of common gram negative bacteria | Blood sample collection beings within 24 to 32 hours of antibiotics administration. Day 1 collections times are zero (predose); 30 minute post dose; 1 hour post dose; 4 hour post dose. Day 2 through 7 collections times occur 2 to 4 hour post dose.
  Number of patients with altered ceftazidime concentrations due to critical illness as measured by less that 50% T>MIC.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bradley, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Childjren's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No